CLINICAL TRIAL: NCT03137758
Title: A Phase I Study of PCUR-101 in Combination With Androgen Suppression Therapy in the Treatment of Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Reformulation of study drug to help reduce the pill burden as higher doses are evaluated.
Sponsor: Pellficure Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCUR101-001
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Level 1 (50 mg) PCUR-101 (Experimental): Starting Dose, 3+3 Cohort Design
  Interventions: Drug: PCUR - 101
- Level 2 (100 mg) PCUR-101 (Experimental)
  Interventions: Drug: PCUR - 101
- Level 3 (150 mg) PCUR-101 (Experimental)
  Interventions: Drug: PCUR - 101
- Level 4 (200 mg) PCUR-101 (Experimental)
  Interventions: Drug: PCUR - 101
- Level 5 (250 mg) PCUR-101 (Experimental)
  Interventions: Drug: PCUR - 101
- Level 6 (300 mg) PCUR-101 (Experimental)
  Interventions: Drug: PCUR - 101

INTERVENTIONS:
Drug: PCUR - 101 — PCUR-101 Capsules 25 mg are solid dosage forms for oral administration

SUMMARY:
This is an open label, non-randomized, Phase I, dose escalation/dose expansion study of PCUR-101 in combination with androgen suppression therapy in the patients with metastatic CRPC

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of metastatic CRPC
* standard of care androgen deprivation treatment
* castrate serum level of testosterone of ≤ 50 ng/dL (≤ 1.73 mmol/L)
* progressive disease while receiving androgen deprivation therapy
* previously treated with abiraterone, enzalutamide alone or in combination AND must have demonstrated evidence of objective progression as per PCWG3 criteria
* adequate hematologic, renal and hepatic function
* KPS of ≥ 70 or ECOG of 0 to 1

Exclusion Criteria:

* pure small cell, neuroendocrine or other variant (non-adenocarcinoma) prostate cancer histology
* use of opiate analgesics for prostate cancer pain within 4 week of treatment start
* more than one sequential second generation AR-directed therapy
* received cytotoxic chemotherapy for either metastatic HSPC or CRPC within the last 12 weeks or other investigational agents within 4 weeks
* history of bleeding disorder
* history of seizure disorder
* concomitant use of therapeutic anticoagulation
* history of or current cardiac issues
* received external beam radiation therapy within 4 weeks
* CTCAE Grade > 2 neuropathy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Toxicities and Adverse Events | 28 days
  determined by type and severity using the most recent version of the CTCAE criteria

SECONDARY OUTCOMES:
Response | up to 2 years
  a combination of the revised RECIST 1.1 criteria and the guidelines for Prostate Cancer Working Group 3 (PCWG3) Criteria
Toxicities and adverse events | up to 2 years
  determined by type and severity using the most recent version of the CTCAE criteria

OTHER OUTCOMES:
Measurement of Serum Cytoine IL-6 | up to 2 years
  Blood based biomarker
Measurement of Urine Polyamines | up to 2 years
  Urine based biomarker

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No